CLINICAL TRIAL: NCT01620372
Title: Constitution d'Une Cohorte Nationale rétrospective de Survivants d'un Cancer Solide de l'Enfant diagnostiqué Avant 2000
Brief Title: French Childhood Cancer Survivor Study
Acronym: FCCSS
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ligue contre le cancer, France (Other); National Research Agency, France (Other); Programme hospitalier de recherche clinique, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: C12-25
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Childhood Solid Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — saliva and blood samples (under another protocol)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Treatment cohort (chemo/radiotherapy): - those who have survived at least 5 years from the date of diagnosis
- Self-questionnaire cohort: - those with a complete address, who come of age, are still alive and sent back a signed consent agreement
- Medical Insurance cohort: - those who come of age and authorize the access to the medical facilities of the French Health Insurance Information System

SUMMARY:
The FCCSS is a multicentric national large-scale collaborative population-based study of children treated for a solid tumor before 2000 in France and before the age of 19 years.

The study is concerned by improving knowledge about the long-term effects caused by cancer and its treatments including adverse health and social outcomes.

The main reason of the FCCSS is to estimate the risk of adverse health and social outcomes that may occur after a cancer treatment and to prevent them by providing adapted follow-up care.

The cohort will be followed for up to 20 years from 2011.

DETAILED DESCRIPTION:
The main objectives of the FCCSS are to:

* estimate the relationship between doses received (radiotherapy, chemotherapy) at a given organ and risk of second malignancy tumors;
* help identify patients at higher risk;
* compare the mortality occurred among the survivors with the general population;
* investigate the consequences of various intensities of exposure to chemotherapy and/or radiation on health outcomes (such as cardiovascular, cerebrovascular and thyroid diseases, diabetes,…);
* characterize survivors with respect to socioeconomic status and quality of life.

The cohort will be ascertained using:

* the medical records from the treatment centers in order to characterize the childhood cancer, estimate doses of radiotherapy received by all organs and measure the chemotherapy administered;
* the French National Identification Registry and the French Death Registry in order to obtain the vital status and the causes of the deaths for the former patients
* a self-questionnaire that covers the entire future of the survivors (e.g. social status, family network, fertile offspring, access to care, access to bank loans, occupation,...);
* the French National Health Insurance Information System that contains data on all reimbursements for health expenditure including medicinal products as well as outpatient medical and nursing care, prescribed or performed by healthcare professionals.

In an initial cohort, we have already studied the iatrogenic effects of the cancer treatments. We have estimated the doses of ionising radiations delivered by radiotherapy to the target volume and by organs at distance. We found an important role of the radiotherapy and chemotherapy in the risk of a second cancer:

* the cancers occuring after childhood cancer are in excess compared to the general population,
* we studied the relationship between the brain radiation dose and the cerebrovascular mortality,
* there is a high risk of cardiac pathology after anthracyclines administration for a childhood cancer,
* cancer treatments increase the risk of second malignant neoplasms in digestive organs after a very long latency period,
* the risk of thyroid adenoma increased with the radiation dose received by the thyroid during childhood cancer treatment, and plateaued at high doses,
* there is a high long-term mortality risk for all types of second malignant neoplasms whatever the treatment received.

ELIGIBILITY:
Inclusion Criteria:

* All types of solid childhood cancer in France
* Age at diagnosis: Below age 19
* Period of diagnosis: between 1st January 1942 and 31st December 1999
* Complete identification (first name, last name, date of birth and place of birth)

Exclusion Criteria:

* Leukaemia cases

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes all types of solid childhood cancer cases (with the exception of leukemia) treated in, or before the end of, 1999.
  The study population is based on the French clinical trials, registries, cohorts and department of paediatric oncology.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2011-11; Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
All health events of interest | by time since diagnosis of solid childhood cancer
  * all causes mortality (e.g. cerebrovascular, cardiovascular,...)
  * all iatrogenic events (e.g. diabetes, thyroid adenomas, cardiac diseases, second malignant solid tumors, secondary leukemia,...)

CONTACTS AND LOCATIONS:
Overall Officials: Florent F. de Vathaire, Ph.D., Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (36):
- France (36):
  - Centre Hospital-Universitaire Hôpital Nord, Amiens
  - Centre Hospitalier-Universitaire, Angers
  - Centre Hospitalier Régional Universitaire Hôpital Saint-Jacques, Besançon
  - Groupe hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Universaitaire Hôpital Côte de Nacre, Caen
  - Centre Hospitalier Universitaire Hôpial Hôtel Dieu, Clermont-Ferrand
  - Centre Hospitalier Universaitaire hôpital d'enfants, Dijon
  - Hôpital La Tronche, Grenoble
  - Centre Oscar Lambret, Lille
  - Hôpital Jeanne De Flandre, Lille
  - Hôpital de la mère et de l'enfant, Limoges
  - Institut d'Hématologie et Oncologie Pédiatrique, Lyon
  - Centre Régional de Lutte Contre le Cancer Centre Léon Bérard, Lyon
  - Hôpital d'Enfants de Margency (HEM) Croix Rouge Française, Margency
  - AP-HM Hôpital de la Timone, Marseille
  - Hôpital Arnaud De Villeneuve, Montpellier
  - Centre Hospitalier Universaitaire Hôpital mère-enfant, Nantes
  - Centre Antoine Lacassagne, Nice
  - GCS Hôpitaux pédiatriques Centre Hospitalier Universitaire Lenval, Nice
  - Institut Curie, Paris
  - Hôpital Armand Trousseau, Paris
  - CHRU de Poitiers La Miletrie, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Universitaire de Reims Hôpital Maison Blanche, Reims
  - Centre Hospitalier Universitaire Hôpital Sud, Rennes
  - Hôpital Charles-Nicolle, Rouen
  - Centre Hospitalier Universitaire Hôpital Nord, Saint-Etienne
  - Centre René Gauducheau de Nantes Atlantique, Saint-Herblain
  - Centre Hospitalier de Saintonge, Saintes
  - Hôpital Hautepierre, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Hôpital des Enfants, Toulouse
  - Hôpital Clocheville, Tours
  - Hôpital Brabois enfants CHU de Nancy, Vandœuvre-lès-Nancy
  - Centre Régional de Lutte Contre le Cancer de Lorraine ALEXIS VAUTRIN, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Pein F, Iserin L, de Vathaire F, Lemerle J. [Cardiac toxicity of cancer treatment regimes in children and adolescents: physiopathology, clinical data and the paediatric oncologist's point of view]. Bull Cancer. 2004 Nov;91 Suppl 3:185-91. French. PMID 15899626
- [Result] Haddy N, El-Fayech C, Guibout C, Adjadj E, Thomas-Teinturier C, Oberlin O, Veres C, Pacquement H, Jackson A, Munzer M, N'Guyen TD, Bondiau PY, Berchery D, Laprie A, Bridier A, Lefkopoulos D, Schlumberger M, Rubino C, Diallo I, de Vathaire F. Thyroid adenomas after solid cancer in childhood. Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):e209-15. doi: 10.1016/j.ijrobp.2012.03.044. Epub 2012 Jun 5. PMID 22672756
- [Result] Tukenova M, Diallo I, Anderson H, Hawkins M, Garwicz S, Sankila R, El Fayech C, Winter D, Rubino C, Adjadj E, Haddy N, Oberlin O, Moller T, Langmark F, Tryggvadottir L, Pacquement H, Svahn-Tapper G, de Vathaire F. Second malignant neoplasms in digestive organs after childhood cancer: a cohort-nested case-control study. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):e383-90. doi: 10.1016/j.ijrobp.2011.05.069. PMID 22284034
- [Result] Haddy N, Mousannif A, Tukenova M, Guibout C, Grill J, Dhermain F, Pacquement H, Oberlin O, El-Fayech C, Rubino C, Thomas-Teinturier C, Le-Deley MC, Hawkins M, Winter D, Chavaudra J, Diallo I, de Vathaire F. Relationship between the brain radiation dose for the treatment of childhood cancer and the risk of long-term cerebrovascular mortality. Brain. 2011 May;134(Pt 5):1362-72. doi: 10.1093/brain/awr071. PMID 21596770
- [Result] Dufour C, Oberlin O, De Vathaire F. [Offspring of childhood cancer survivors]. Arch Pediatr. 2010 Jun;17(6):926-7. doi: 10.1016/S0929-693X(10)70182-2. No abstract available. French. PMID 20654964
- [Result] Tukenova M, Guibout C, Hawkins M, Quiniou E, Mousannif A, Pacquement H, Winter D, Bridier A, Lefkopoulos D, Oberlin O, Diallo I, de Vathaire F. Radiation therapy and late mortality from second sarcoma, carcinoma, and hematological malignancies after a solid cancer in childhood. Int J Radiat Oncol Biol Phys. 2011 Jun 1;80(2):339-46. doi: 10.1016/j.ijrobp.2010.02.004. Epub 2010 Jun 18. PMID 20646844
- [Result] Tukenova M, Diallo I, Hawkins M, Guibout C, Quiniou E, Pacquement H, Dhermain F, Shamsaldin A, Oberlin O, de Vathaire F. Long-term mortality from second malignant neoplasms in 5-year survivors of solid childhood tumors: temporal pattern of risk according to type of treatment. Cancer Epidemiol Biomarkers Prev. 2010 Mar;19(3):707-15. doi: 10.1158/1055-9965.EPI-09-1156. Epub 2010 Mar 3. PMID 20200431
- [Result] Tukenova M, Guibout C, Oberlin O, Doyon F, Mousannif A, Haddy N, Guerin S, Pacquement H, Aouba A, Hawkins M, Winter D, Bourhis J, Lefkopoulos D, Diallo I, de Vathaire F. Role of cancer treatment in long-term overall and cardiovascular mortality after childhood cancer. J Clin Oncol. 2010 Mar 10;28(8):1308-15. doi: 10.1200/JCO.2008.20.2267. Epub 2010 Feb 8. PMID 20142603
- [Result] Diallo I, Haddy N, Adjadj E, Samand A, Quiniou E, Chavaudra J, Alziar I, Perret N, Guerin S, Lefkopoulos D, de Vathaire F. Frequency distribution of second solid cancer locations in relation to the irradiated volume among 115 patients treated for childhood cancer. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):876-83. doi: 10.1016/j.ijrobp.2009.01.040. Epub 2009 Apr 20. PMID 19386434
- [Result] Nguyen F, Rubino C, Guerin S, Diallo I, Samand A, Hawkins M, Oberlin O, Lefkopoulos D, De Vathaire F. Risk of a second malignant neoplasm after cancer in childhood treated with radiotherapy: correlation with the integral dose restricted to the irradiated fields. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):908-15. doi: 10.1016/j.ijrobp.2007.10.034. PMID 18262102
- [Result] Guerin S, Hawkins M, Shamsaldin A, Guibout C, Diallo I, Oberlin O, Brugieres L, de Vathaire F. Treatment-adjusted predisposition to second malignant neoplasms after a solid cancer in childhood: a case-control study. J Clin Oncol. 2007 Jul 1;25(19):2833-9. doi: 10.1200/JCO.2006.09.6719. PMID 17602088
- [Result] Guerin S, Guibout C, Shamsaldin A, Dondon MG, Diallo I, Hawkins M, Oberlin O, Hartmann O, Michon J, Le Deley MC, de Vathaire F. Concomitant chemo-radiotherapy and local dose of radiation as risk factors for second malignant neoplasms after solid cancer in childhood: a case-control study. Int J Cancer. 2007 Jan 1;120(1):96-102. doi: 10.1002/ijc.22197. PMID 17013899
- [Result] Haddy N, Le Deley MC, Samand A, Diallo I, Guerin S, Guibout C, Oberlin O, Hawkins M, Zucker JM, de Vathaire F. Role of radiotherapy and chemotherapy in the risk of secondary leukaemia after a solid tumour in childhood. Eur J Cancer. 2006 Nov;42(16):2757-64. doi: 10.1016/j.ejca.2006.05.034. Epub 2006 Sep 11. PMID 16965909
- [Result] Guibout C, Adjadj E, Rubino C, Shamsaldin A, Grimaud E, Hawkins M, Mathieu MC, Oberlin O, Zucker JM, Panis X, Lagrange JL, Daly-Schveitzer N, Chavaudra J, de Vathaire F. Malignant breast tumors after radiotherapy for a first cancer during childhood. J Clin Oncol. 2005 Jan 1;23(1):197-204. doi: 10.1200/JCO.2005.06.225. PMID 15625374
- [Result] Menu-Branthomme A, Rubino C, Shamsaldin A, Hawkins MM, Grimaud E, Dondon MG, Hardiman C, Vassal G, Campbell S, Panis X, Daly-Schveitzer N, Lagrange JL, Zucker JM, Chavaudra J, Hartman O, de Vathaire F. Radiation dose, chemotherapy and risk of soft tissue sarcoma after solid tumours during childhood. Int J Cancer. 2004 May 20;110(1):87-93. doi: 10.1002/ijc.20002. PMID 15054872
- [Result] Rubino C, Adjadj E, Guerin S, Guibout C, Shamsaldin A, Dondon MG, Valteau-Couanet D, Hartmann O, Hawkins M, de Vathaire F. Long-term risk of second malignant neoplasms after neuroblastoma in childhood: role of treatment. Int J Cancer. 2003 Dec 10;107(5):791-6. doi: 10.1002/ijc.11455. PMID 14566829
- [Result] Guerin S, Dupuy A, Anderson H, Shamsaldin A, Svahn-Tapper G, Moller T, Quiniou E, Garwicz S, Hawkins M, Avril MF, Oberlin O, Chavaudra J, de Vathaire F. Radiation dose as a risk factor for malignant melanoma following childhood cancer. Eur J Cancer. 2003 Nov;39(16):2379-86. doi: 10.1016/s0959-8049(03)00663-4. PMID 14556931
- [Result] de Vathaire F, Hardiman C, Shamsaldin A, Campbell S, Grimaud E, Hawkins M, Raquin M, Oberlin O, Diallo I, Zucker JM, Panis X, Lagrange JL, Daly-Schveitzer N, Lemerle J, Chavaudra J, Schlumberger M, Bonaiti C. Thyroid carcinomas after irradiation for a first cancer during childhood. Arch Intern Med. 1999 Dec 13-27;159(22):2713-9. doi: 10.1001/archinte.159.22.2713. PMID 10597762
- [Result] de Vathaire F, Hawkins M, Campbell S, Oberlin O, Raquin MA, Schlienger JY, Shamsaldin A, Diallo I, Bell J, Grimaud E, Hardiman C, Lagrange JL, Daly-Schveitzer N, Panis X, Zucker JM, Sancho-Garnier H, Eschwege F, Chavaudra J, Lemerle J. Second malignant neoplasms after a first cancer in childhood: temporal pattern of risk according to type of treatment. Br J Cancer. 1999 Apr;79(11-12):1884-93. doi: 10.1038/sj.bjc.6690300. PMID 10206309
- [Result] Little MP, de Vathaire F, Shamsaldin A, Oberlin O, Campbell S, Grimaud E, Chavaudra J, Haylock RG, Muirhead CR. Risks of brain tumour following treatment for cancer in childhood: modification by genetic factors, radiotherapy and chemotherapy. Int J Cancer. 1998 Oct 29;78(3):269-75. doi: 10.1002/(SICI)1097-0215(19981029)78:33.0.CO;2-T. PMID 9766556
- [Result] Le Vu B, de Vathaire F, Shamsaldin A, Hawkins MM, Grimaud E, Hardiman C, Diallo I, Vassal G, Bessa E, Campbell S, Panis X, Daly-Schveitzer N, Lagrange JL, Zucker JM, Eschwege F, Chavaudra J, Lemerle J. Radiation dose, chemotherapy and risk of osteosarcoma after solid tumours during childhood. Int J Cancer. 1998 Jul 29;77(3):370-7. doi: 10.1002/(sici)1097-0215(19980729)77:33.0.co;2-c. PMID 9663598
- [Result] de Vathaire F, Shamsaldin A, Grimaud E, Campbell S, Guerra M, Raquin M, Bessa E, Hardiman C, Jan P, Rumeau N, et al. Solid malignant neoplasms after childhood irradiation: decrease of the relative risk with time after irradiation. C R Acad Sci III. 1995 Apr;318(4):483-90. PMID 7648361
- [Result] Pein F, Sakiroglu O, Dahan M, Lebidois J, Merlet P, Shamsaldin A, Villain E, de Vathaire F, Sidi D, Hartmann O. Cardiac abnormalities 15 years and more after adriamycin therapy in 229 childhood survivors of a solid tumour at the Institut Gustave Roussy. Br J Cancer. 2004 Jul 5;91(1):37-44. doi: 10.1038/sj.bjc.6601904. PMID 15162142
- [Result] Guldner L, Haddy N, Pein F, Diallo I, Shamsaldin A, Dahan M, Lebidois J, Merlet P, Villain E, Sidi D, Sakiroglu O, Hartmann O, Leftakopoulos D, de Vathaire F. Radiation dose and long term risk of cardiac pathology following radiotherapy and anthracyclin for a childhood cancer. Radiother Oncol. 2006 Oct;81(1):47-56. doi: 10.1016/j.radonc.2006.08.020. Epub 2006 Sep 20. PMID 16989913
- [Result] Shamsaldin A, Grimaud E, Hardiman C, Diallo I, de-Vathaire F, Chavaudra J. Dose distribution throughout the body from radiotherapy for Hodgkin's disease in childhood. Radiother Oncol. 1998 Oct;49(1):85-90. doi: 10.1016/s0167-8140(98)00110-8. PMID 9886702
- [Result] de Vathaire F, Francois P, Schlumberger M, Schweisguth O, Hardiman C, Grimaud E, Oberlin O, Hill C, Lemerle J, Flamant R. Epidemiological evidence for a common mechanism for neuroblastoma and differentiated thyroid tumour. Br J Cancer. 1992 Mar;65(3):425-8. doi: 10.1038/bjc.1992.87. PMID 1558799
- [Result] de Vathaire F, Francois P, Hill C, Schweisguth O, Rodary C, Sarrazin D, Oberlin O, Beurtheret C, Dutreix A, Flamant R. Role of radiotherapy and chemotherapy in the risk of second malignant neoplasms after cancer in childhood. Br J Cancer. 1989 May;59(5):792-6. doi: 10.1038/bjc.1989.165. PMID 2736215
- [Result] de Vathaire F, Schweisguth O, Rodary C, Francois P, Sarrazin D, Oberlin O, Hill C, Raquin MA, Dutreix A, Flamant R. Long-term risk of second malignant neoplasm after a cancer in childhood. Br J Cancer. 1989 Mar;59(3):448-52. doi: 10.1038/bjc.1989.92. PMID 2930714
- [Result] de Vathaire F, Francois P, Schweisguth O, Oberlin O, Le MG. Irradiated neuroblastoma in childhood as potential risk factor for subsequent thyroid tumour. Lancet. 1988 Aug 20;2(8608):455. doi: 10.1016/s0140-6736(88)90445-x. No abstract available. PMID 2900383
- [Result] de Vathaire F, El-Fayech C, Ben Ayed FF, Haddy N, Guibout C, Winter D, Thomas-Teinturier C, Veres C, Jackson A, Pacquement H, Schlumberger M, Hawkins M, Diallo I, Oberlin O. Radiation dose to the pancreas and risk of diabetes mellitus in childhood cancer survivors: a retrospective cohort study. Lancet Oncol. 2012 Oct;13(10):1002-10. doi: 10.1016/S1470-2045(12)70323-6. Epub 2012 Aug 23. PMID 22921663
- [Derived] de Vathaire F, Haddy N, Allodji RS, Hawkins M, Guibout C, El-Fayech C, Teinturier C, Oberlin O, Pacquement H, Diop F, Kalhouche A, Benadjaoud M, Winter D, Jackson A, Bezin Mai-Quynh G, Benabdennebi A, Llanas D, Veres C, Munzer M, Nguyen TD, Bondiau PY, Berchery D, Laprie A, Deutsch E, Lefkopoulos D, Schlumberger M, Diallo I, Rubino C. Thyroid Radiation Dose and Other Risk Factors of Thyroid Carcinoma Following Childhood Cancer. J Clin Endocrinol Metab. 2015 Nov;100(11):4282-90. doi: 10.1210/jc.2015-1690. Epub 2015 Sep 1. PMID 26327481
- See also: Center for research in epidemiology and population Health - U1018 Inserm — http://cesp.inserm.fr/en/